CLINICAL TRIAL: NCT03799588
Title: Transmitted Lung Pressure Values With Biphasic Chest Cuirass
Brief Title: Transmitted Lung Pressures With Biphasic Chest Cuirass
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: personnel have left the facility
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Bree Cyrene Kramer, Assistant Clinical Professor of Pediatrics, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00002374
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Lung Diseases
Keywords: Pediatrics; biphasic chest cuirass; transpulmonary pressure
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: After routine intubation for elective urologic procedures in the OR, the patient will be placed on a biphasic chest cuirass after anesthesia induction. A esophageal manometer will then be placed to measure transpulmonary pressures. The patient will be switched off the anesthesia ventilator and the biphasic chest cuirass will begin negative pressure ventilation. During this time, the patient will continue to receive inhalation anesthetic gas. After 30 minutes, the biphasic chest cuirass will terminate and the patient will again receive positive pressure ventilation via the anesthesia ventilator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biphasic Chest Cuirass Arm (Experimental): This is the only arm in the study and all patients will receive negative pressure ventilation via the biphasic chest cuirass.
  Interventions: Device: Biphasic Chest Cuirass

INTERVENTIONS:
Device: Biphasic Chest Cuirass — Patients will have a esophageal manometer placed after intubation and before initiation of negative pressure ventilation.

SUMMARY:
This study will examine the correlation between the transpulmonary pressure and the actual setting on the biphasic chest cuirass device is the primary study end point.

DETAILED DESCRIPTION:
Conventional mechanical ventilation is known as positive pressure ventilation (PPV) because the machine delivers positive pressure directly into the airways to ventilate and expand the lungs. In a healthy lung, inflation occurs when the pressure inside the lung is greater than the pressure outside the lung. This transpulmonary pressure is the difference between the pressure inside the lung (in the alveolus) and the pressure just outside the lung (the pleural cavity). Since positive pressure ventilation delivers pressure directly into the airways, the transpulmonary pressure is increased by making the lung pressure more positive. This is markedly different than physiologic breathing and carries an increased risk of ventilator-associated lung injury1. In the setting of sick lungs, where the pressure required to open collapsed areas of lung may be more than areas of healthy lung, this higher pressure can in turn cause damage to the areas of healthy lung. The known effects of this ventilator-associated lung injury from positive pressure ventilation can be avoided with the use of negative pressure ventilation. In negative pressure ventilation (NPV), the transpulmonary pressure is increased by making the pleural pressure more negative. This is achieved by using a plastic shell that covers the chest and generates negative pressure between the plastic shell and the chest. This pressure is distributed more evenly across a large surface of the chest wall and results in more uniform lung expansion. As a result, NPV results in better oxygen delivery and less lung injury than positive pressure ventilation2.

However, despite the extensive use of NPV in other countries, there is little data available regarding the transpulmonary pressure that these machines can generate; i.e. how well does negative pressure in the plastic shell transmit to the pleural cavity to expand the lung. There is a large amount of data supporting the use of biphasic cuirass ventilation to minimize lung damage3 and improve hemodynamics4-9, but no studies have been done to date that look at the transpulmonary pressure and how it differs depending on age and size. It is still unclear what optimal pressure is required via the chest cuirass to expand and ventilate the lungs via. It is also unknown what maximum pressures can be used before the lung becomes overinflated and complications arise.

This study will examine the correlation between the transpulmonary pressure and the actual setting on the biphasic chest cuirass device is the primary study end point.

ELIGIBILITY:
Inclusion Criteria:

1. Are between the age of 6 months and 5 years
2. Undergo circumcision, hypospadias repair, or orchidopexy in the operating room of the John R. Oishei Children's Hospital

Exclusion Criteria:

1. Previous history of chronic lung disease or cyanotic heart disease or
2. Patients with significant chest wall abnormalities or other abnormalities that preclude proper placement of the biphasic chest cuirass.

Ages: 6 Months to 5 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Transpulmonary Pressure Deliverance | 1 year
  Examining the correlation between the transpulmonary pressure and the actual setting on the biphasic chest cuirass device is the primary study end point.

CONTACTS AND LOCATIONS:
Overall Officials: Bree C Kramer, DO, Principal Investigator — University at Buffalo
Locations (1):
- Oishei Children's Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scholz SE, Knothe C, Thiel A, Hempelmann G. Improved oxygen delivery by positive pressure ventilation with continuous negative external chest pressure. Lancet. 1997 May 3;349(9061):1295-6. doi: 10.1016/S0140-6736(05)62507-X. No abstract available. PMID 9142069
- [Background] Petros AJ, Fernando SS, Shenoy VS, al-Saady NM. The Hayek oscillator. Nomograms for tidal volume and minute ventilation using external high frequency oscillation. Anaesthesia. 1995 Jul;50(7):601-6. doi: 10.1111/j.1365-2044.1995.tb15112.x. PMID 7653758